CLINICAL TRIAL: NCT03005938
Title: Influence of the Spinal Manipulation on Muscle Spasticity and Manual Dexterity in Children With Cerebral Palsy, Randomized Control Trial.
Brief Title: Influence of the Spinal Manipulation on Muscle Spasticity and Manual Dexterity in Cerebral Palsy.
Acronym: SpiManCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Clinic of Rehabilitation, Ukraine (Other)
Responsible Party: Principal Investigator, Oleh Kachmar, Head of Innovative Technologies Department, International Clinic of Rehabilitation, Ukraine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: N-09-2016
Record Dates: First submitted 2016-12-21; First posted 2016-12-30 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral Palsy; Spinal Manipulation; Muscle Spasticity; Manual Dexterity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal manipulation (Experimental): Spinal manipulation
  Interventions: Procedure: Spinal manipulation
- Imitation of the spinal manipulation (Sham Comparator): Imitation of the spinal manipulation
  Interventions: Procedure: Imitation of the spinal manipulation

INTERVENTIONS:
Procedure: Spinal manipulation — Spinal manipulation (SM) is a therapeutic intervention performed on spinal articulations in which force is applied to the spine. The selected joint is moved to its end range of motion, followed by application of an rapid impulse or thrust to achieve a gapping of the target joint.
  SM is performed by an orthopedic medical doctor certified in Manual Therapy. After manual evaluation, high-velocity low-amplitude SM is carried out in all regions of the spine, including thoracic adjustments in the prone position, lumbar manipulation in lateral recumbent position, and cervical manipulation in sitting position.
  Other Names: Biomechanical correction of the spine
  Arms: Spinal manipulation
Procedure: Imitation of the spinal manipulation — Imitation of the SM physically and visually resembles the act of SM. It comprises placing the patient in the same positions and performing the same movements as during SM but without applying the force in the end range of motion.
  Other Names: Sham manipulation
  Arms: Imitation of the spinal manipulation

SUMMARY:
The aim of the study is to evaluate a short term influence of the Spinal Manipulation (SM) on the wrist muscles spasticity and manual dexterity in children with spastic Cerebral Palsy.

Effect of SM and imitation of the SM has to be compared in the double-blinded randomized clinical trial.

DETAILED DESCRIPTION:
Muscle spasticity is an important clinical syndrome of Cerebral Palsy (CP) resulting from upper motor neuron lesion, and its reduction is a significant therapeutic target for optimizing motor performance.

Investigator's recent study describes decrease in spasticity after SM in a group of children with CP. But that case series has no control group and the sample size was small so it does not prove the influence of the SM on the muscle spasticity.

The purpose of the present study is to evaluate influence of the SM on muscle spasticity and on manual dexterity of the child with CP in a double-blind randomized clinical trial with two arms: SM (experimental group) and imitation of SM (control group).

Children admitted to the International Clinic of Rehabilitation are selected according to inclusion-exclusion criteria and invited to participate. After getting the permission the baseline assessment is performed.

Patients are allocated to the experimental or control group using stratified randomization. Medical doctor certified in Manual Therapy performs the intervention (SM in the experimental group and imitation in the control group) and in 15 minutes the second assessment is performed. Investigators, children and parents are blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Spastic uni-, bilateral Cerebral Palsy
* Manual Ability classification level (MACS) - I-III level
* Modified Ashworth scale (MAS) grade 1-3 in wrist or fingers flexors

Exclusion Criteria:

* Dyskinetic or ataxic syndrome
* Less than 40 degrees of passive wrist extension with fingers extended
* Botox injections in hand muscles during last year or recent antispastic drugs
* Fracture in hand or forearm less than 6 month prior to examination
* Uncooperative behavior, inability to understand and comply with instructions
* Severe pain preventing the child from being able to complete examinations

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Change of muscle spasticity after the intervention | Baseline assesment and 15 min after intervention
  Quantitative, instrumental spasticity measurement is preformed using the Neuroflexor device. It is measuring resistance to passive movements of the wrist performed with different speed and calculates components of muscle tone, separating spasticity as reflex phenomenon from resistance due to secondary changes of the muscles and tendons.

SECONDARY OUTCOMES:
Change of manual dexterity after the intervention | Baseline assesment and 15 min after intervention
  Manual dexterity is evaluated using Box and Blocks test. The score is the number of blocks carried by hand from one compartment to the other in one minute.

CONTACTS AND LOCATIONS:
Overall Officials: Oleh Kachmar, MD, PhD, Principal Investigator — International Clinic of Rehabilitation, Ukraine
Locations (1):
- International Clinic of Rehabilitation, Truskavets, Lviv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kachmar O, Voloshyn T, Hordiyevych M. Changes in Muscle Spasticity in Patients With Cerebral Palsy After Spinal Manipulation: Case Series. J Chiropr Med. 2016 Dec;15(4):299-304. doi: 10.1016/j.jcm.2016.07.003. Epub 2016 Sep 28. PMID 27857638
- [Background] Lindberg PG, Gaverth J, Islam M, Fagergren A, Borg J, Forssberg H. Validation of a new biomechanical model to measure muscle tone in spastic muscles. Neurorehabil Neural Repair. 2011 Sep;25(7):617-25. doi: 10.1177/1545968311403494. Epub 2011 Apr 13. PMID 21490269
- [Background] Koziavkin VI, Kachmar OA, Voloshin TB, Gordievich MS. [Components of the muscle tone and quantitative spasticity measurement technique]. The Journal of Neuroscience of B. M. Mankovsky. 2015, vol.3,N1:72-76. in Ukrainian.